CLINICAL TRIAL: NCT03496636
Title: Autologous Ovarian Tissue Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050305
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Female Infertility
Keywords: Ovary; Transplant
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ovarian tissue transplant (Experimental): Transplantation of ovarian tissue into the abdomen. Only for patients who have previously frozen ovarian tissue
  Interventions: Procedure: Ovarian tissue transplant

INTERVENTIONS:
Procedure: Ovarian tissue transplant — Pieces of previously frozen ovarian cortex will be put in the abdomen laparoscopically, or with mini laparotomy

SUMMARY:
Chemotherapy and radiation for cancer and other conditions can cause infertility. Several centers around the world are cryopreserving ovarian tissue from these patients though an experimental protocol, including the Fertility Preservation Program in Pittsburgh (protocol PRO08050491). The objective of this study is to study the efficacy and safety of autologous tissue transplantation in patients diagnosed with primary ovarian insufficiency after chemotherapy and/or radiation treatments.

DETAILED DESCRIPTION:
This investigation involves patient enrollment, thaw and surgical transplantation of previously collected cryopreserved ovarian cortical tissue, a series of follow-up assessments during the first 2 years after transplantation and an annual survey after year 2.

Screening visit (standard fertility consultation):

1. The subject will complete a medical and reproductive history to document menstrual function and suitability for pregnancy.
2. The subject will have standard fertility testing (including but not limited to serum Follicle Stimulating Hormone (FSH), Estradiol (E2), and Anti-Mullerian Hormone (AMH), luteinizing hormone (LH), testosterone and progesterone).
3. Vaginal ultrasound will be performed for measures of ovarian volume and antral follicle counts.
4. A pregnancy test will be performed to rule out pregnancy.
5. Each potential subject will undergo a comprehensive fertility consult including counseling regarding the extent to which participation in this study might be of ultimate benefit. Alternatives to participation include: continuing to try to conceive on her own, use of donor oocytes or embryos, or adoption.
6. The subject will have to obtain clearance from her oncologist and will be counseled by a reproductive endocrinologist to determine whether she is healthy enough to consider pregnancy and to discuss the potential risks and benefits of the study.

Visit #1 - pre-op visit (can be combined with initial screening visit):

Eligible subjects will be consented by the study physician and complete the same infectious disease testing as was performed at the time of ovarian tissue freezing (including but not limited to HIV 1&2, HTLV 1&2, Hepatitis B, Hepatitis C, syphilis, chlamydia, gonorrhea, CMV, West Nile virus). The subjects will also complete Fertility quality of life survey (FertiQoL). FertiQoL is a validated measure of quality of life in people experiencing fertility problems.

Only after confirming eligibility, obtaining informed consent and completing baseline measures, ovarian tissue thawing and transplantation will be performed.

Visit #2 - Ovarian tissue transplantation:

At the time of ovarian tissue thawing, an outpatient laparoscopy (or minilaparotomy if the patient is not deemed to be a good candidate for laparoscopic surgery) will be performed under general anesthesia. Ovarian cortical tissue will be transplanted within the pelvis according to the most effective available techniques.

Visit #3: Post-operative assessment:

Within six weeks of transplant, a postoperative follow-up assessment will be conducted to ensure adequate patient recovery and emotional well-being. Blood tests (including but not limited to serum FSH, E2, and AMH, LH, testosterone and progesterone), pelvic ultrasound and FertiQoL survey, will be conducted to assess reproductive hormone levels, menstrual function, complications from surgery, pregnancy, medical and medication history, and cancer relapse. Referral to the clinical counselor may be made, if indicated.

Visits #4, #5, #6, #7 and #8 at 3, 6, 9, 12 and 24 months post-op:

A series of 5 additional follow-up assessments will be conducted during the first 2 years after transplant with Reproductive Endocrinology and Infertility to assess reproductive hormone levels, menstrual function, complications from surgery, pregnancy, changes in medical and medication status, and cancer relapse. A visit may be added at the time menstruation is restored if this occurs between regularly scheduled visits. At each follow up visit hormone testing is performed, vaginal ultrasound and FertiQoL survey will be administered. Additional clinical follow-up and testing may be determined in consultation with the subject's oncologist.

Annual Survey:

Starting year 3 post-transplantation, each subject will be surveyed annually. The survey is voluntary and confidential and will be conducted by scripted phone interview or self-administered survey through secure email. The survey will include questions about menstrual/pregnancy history, new diagnoses or treatments, and feelings about participating in the study. Detailed information about pregnancy and birth outcomes will be collected by a combination of survey and chart review. Outcome data including remission, relapse or death, will be collected. Contact information will also be updated.

ELIGIBILITY:
Inclusion Criteria:

* Previously cryopreserved ovarian tissue
* Ovarian insufficiency and/or candidate for pregnancy
* Good health
* Oncologist's clearance

Exclusion Criteria:

* Patients considered to be high risk for surgical complications
* Women with contraindication for pregnancy if goal is to achieve pregnancy
* Women positive for the BRCA mutations
* Women with a history of leukemia, ovarian cancer or a cancer that likely involved ovaries at the time of ovarian tissue collection
* Women with psychological, psychiatric, or other conditions which prevent giving fully informed consent
* Current pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in reproductive hormone levels after ovarian tissue transplant | 1,3,6,9,12 and 24 months post-transplantation
  Measure of reproductive hormone levels (FSH, AMH, LH E2 and others) to detect graft function
Return of regular monthly menstrual cycles | Through study completion, up to 15 years
  Onset of regular monthly menstrual cycles after transplantation would indicate graft function. This needs to be analyzed at multiple time points to assess if regular monthly menstrual cycles have ceased, which could indicate graft failure.
Achievement of successful pregnancy, measured by live birth | Through study completion, up to 15 years
  Indicates recovery of ovarian function

SECONDARY OUTCOMES:
Cancer recurrence as determined by patient's oncologist | Through study completion, up to 15 years
  Indicates cancer recurrence
Surgical complications of ovarian tissue transplantation | 1,3,6,9,12 and 24 months post-transplantation
  Infection, hospital readmission, re-operation
Fertility quality of life (FertiQoL) survey results | 1,3,6,9,12 and 24 months post-transplantation
  Measure quality of life in individuals experiencing fertility problems

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish individual participant data. The investigators will also report each individual participants data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: We will share IPD with the patient (and only the patient) within one year of enrollment. We share study protocol and ICF with collaborating sites upon request. De-identified IDP is shared with collaborating sites annually.
Access Criteria: De-identified research data will be shared with collaborators via e-mail, and with the broader scientific community via publication and presentations at national/international meetings.